CLINICAL TRIAL: NCT03627273
Title: Comparison of 6 Minute Walk Test With and Without Walker
Brief Title: 6MWT With and Without Walker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 6MWTrollator
Record Dates: First submitted 2018-07-15; First posted 2018-08-13 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Healthy; Elderly

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- walker (Experimental): '6 minutes walking test' with a walker
  Interventions: Diagnostic Test: 6 minutes walking test with walker
- no walker (Active Comparator): '6 minutes walking test' without walker
  Interventions: Diagnostic Test: 6 minutes walking test

INTERVENTIONS:
Diagnostic Test: 6 minutes walking test with walker — to walk during 6 minutes with walker
  Arms: walker
Diagnostic Test: 6 minutes walking test — to walk during 6 minutes with walker
  Arms: no walker

SUMMARY:
Elderly subjects repeated 6MWT with or without walker

ELIGIBILITY:
Inclusion Criteria:

* clinically stable
* aged over 65 years
* could walk
* did not use walker frames in routine

Exclusion Criteria:

* criteria outlined in the European respiratory society/American thoracic society technical standard related to 6MWT
* impaired cognitive function

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 86 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
six minutes walking test | six minutes
  distance

SECONDARY OUTCOMES:
Modified Borg scale | six minutes
  dyspnea
heart rate | six minutes
  heart beat rate
pulsed oxygen saturation | six minutes
  saturation pulsed oxygen

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No